CLINICAL TRIAL: NCT06619145
Title: Oliceridine for Analgesia After Cardiac Surgery
Brief Title: 1.Comparison of the Analgesic Effect of Remifentanil Group and Different Dose Groups of Oliceridine in Postoperative Patients Undergoing Cardiac Surgery 2.Exploring the Hemodynamic Effects of Analgesic Regimens With Different Doses of Oliceridine After Cardiac Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20240924-07
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Oliceridine; Postoperative Cardiac Surgery
MeSH Terms: interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remifentanil (No Intervention)
- High dose Oliceridine (Experimental): High dose Oliceridine
  Interventions: Drug: High dose Oliceridine
- Low dose Oliceridine (Experimental): Low dose Oliceridine
  Interventions: Drug: Low dose Oliceridine

INTERVENTIONS:
Drug: Low dose Oliceridine — Low dose Oliceridine
  Arms: Low dose Oliceridine
Drug: High dose Oliceridine — High dose Oliceridine
  Arms: High dose Oliceridine

SUMMARY:
Cardiac surgery has the characteristics of long duration and large amount of intraoperative bleeding, easy to involve multiple organs and severe tissue injury, which is one of the most serious surgical procedures with postoperative pain and the incidence of postoperative pain after open-heart surgery is as high as 50%, with the incidence of moderate-to-severe pain ranging from 3% to 18% . Currently, opioids are commonly used in clinical practice for postoperative cardiac analgesia, but due to the abnormal cardiac structure of cardiac surgery patients, surgery and extracorporeal circulation effects, hemodynamic fluctuations and respiratory depression, nausea and vomiting, dizziness, constipation, and other adverse reactions occur during analgesia [3]. Therefore, it is especially necessary to find an analgesic drug with good analgesic effect and able to reduce such adverse effects.

Oliceridine is a G-protein biased μ-opioid receptor agonist, which selectively activates the G-protein signaling pathway and significantly reduces the activation of the β-inhibitory protein pathway, preserving the analgesic effect while reducing the opioid-related adverse effects, and is currently used for intraoperative analgesia and analgesic treatment of acute moderate-to-severe pain occurring after surgery such as abdominal surgery and bunion bursitis, and is mostly administered by a single injection into the vein .A series of national and international clinical studies have been conducted on OliceridineA phase 1 clinical trial study conducted by Soergel et al. demonstrated that in healthy subjects, 3 and 4.5 mg ofOliceridine demonstrated higher peak analgesia (75 sec latency) compared to morphine. In addition, all doses were associated with lower respiratory drive reductions compared to morphine (- 7.3, - 7.6, and - 9.4 h*L/min vs - 15.9 h*L/min). Respiratory depression persisted with Oliceridine but was very transient, and subjects on the 1.5 mg and 3 mg doses experienced less nausea compared to subjects on the 4.5 mg dose and morphine. Overall, the 3 mg dose provided significant efficacy while still maintaining the reduction in PONV demonstrated by the low dose of choline.

To further investigate the effects of Oliceridine on the respiratory system, Simons et al. conducted a crossover study of 18 healthy elderly volunteers. The study found that while low doses of Oliceridine did not result in any significant respiratory effects, high doses of Oliceridine and two doses of morphine resulted in respiratory depression that peaked 0.5 to 1 hour after administration. However, similar to the earlier findings of Soergel et al, the respiratory depression induced by Oliceridine was more transient, characterized by a more rapid return to baseline, with an equilibrium half-life at the blood effector site of 44.3 ± 6.1 minutes compared with 214 ± 27 minutes for morphine.A subsequent phase III study was also conducted on the use of Oliceridine in the management of moderate to severe acute postoperative pain after abdominoplasty. The results showed that Oliceridine is a safe and effective intravenous analgesic for the relief of moderate to severe acute postoperative pain in patients undergoing abdominoplasty. Since the low-dose regimen of 0.1 mg of oseltamivirine was superior to placebo but not as effective as the morphine regimen, safety comparisons with morphine were only relevant to the 2 isoanalgesic dose groups of 0.35 and 0.5 mg, and oseltamivirine showed a favorable safety profile in terms of respiratory and gastrointestinal adverse effects tolerability compared with morphine. This suggests that Oliceridine may offer a new therapeutic option for patients with moderate to severe acute pain requiring intravenous opioids.Based on the relatively long duration of analgesia in postoperative cardiac surgery patients, there is a need to explore drugs with the advantages of better analgesic effect, less hemodynamic impact, sustained analgesia with fewer adverse effects, and rapid metabolism after discontinuation of the drug. Combining the existing research base of this project and the above domestic and international findings, we propose the conjecture that Oliceridine may provide better analgesia with fewer adverse effects in the postoperative period of cardiac surgery relative to other opioid analgesic drugs. In this study, we propose to study the analgesic effect of different doses of Oliceridine for pumping in postoperative cardiac surgery patients, its effect on hemodynamics and safety assessment, and we intend to expect to determine the optimal dosing regimen for postoperative cardiac analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative patients undergoing cardiac surgery from November 2024 to October 2025

Exclusion Criteria:

* body mass index (BMI) > 35 kg/m2 or weight < 40 kg; ② age < 18 years old, or ≥ 80 years old; ③ sleep apnea; ④ opioid allergy; ⑤ use of analgesic drugs for chronic pain; ⑥ prolongation of the Q-T interval; ⑦ serious dysfunction of the liver and kidneys and other organs; ⑧ the presence of postoperative low cardiac output, hemorrhage, vascular paralysis syndrome, etc. Causes circulatory disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
CPOT score | 15 minutes, 30 minutes, 1 hour (h), 4 h, 8 h, 12 h, 24 hours (h) after loading dose drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singla NK, Skobieranda F, Soergel DG, Salamea M, Burt DA, Demitrack MA, Viscusi ER. APOLLO-2: A Randomized, Placebo and Active-Controlled Phase III Study Investigating Oliceridine (TRV130), a G Protein-Biased Ligand at the mu-Opioid Receptor, for Management of Moderate to Severe Acute Pain Following Abdominoplasty. Pain Pract. 2019 Sep;19(7):715-731. doi: 10.1111/papr.12801. Epub 2019 Jun 24. PMID 31162798
- [Result] Viscusi ER, Webster L, Kuss M, Daniels S, Bolognese JA, Zuckerman S, Soergel DG, Subach RA, Cook E, Skobieranda F. A randomized, phase 2 study investigating TRV130, a biased ligand of the mu-opioid receptor, for the intravenous treatment of acute pain. Pain. 2016 Jan;157(1):264-272. doi: 10.1097/j.pain.0000000000000363. PMID 26683109
- [Result] Dahan A, van Dam CJ, Niesters M, van Velzen M, Fossler MJ, Demitrack MA, Olofsen E. Benefit and Risk Evaluation of Biased mu-Receptor Agonist Oliceridine versus Morphine. Anesthesiology. 2020 Sep;133(3):559-568. doi: 10.1097/ALN.0000000000003441. PMID 32788558
- [Result] Soergel DG, Subach RA, Burnham N, Lark MW, James IE, Sadler BM, Skobieranda F, Violin JD, Webster LR. Biased agonism of the mu-opioid receptor by TRV130 increases analgesia and reduces on-target adverse effects versus morphine: A randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Pain. 2014 Sep;155(9):1829-1835. doi: 10.1016/j.pain.2014.06.011. Epub 2014 Jun 19. PMID 24954166
- [Result] Nafziger AN, Arscott KA, Cochrane K, Skobieranda F, Burt DA, Fossler MJ. The Influence of Renal or Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of Oliceridine. Clin Pharmacol Drug Dev. 2020 Jul;9(5):639-650. doi: 10.1002/cpdd.750. Epub 2019 Nov 7. PMID 31697049
- [Result] Viscusi ER, Skobieranda F, Soergel DG, Cook E, Burt DA, Singla N. APOLLO-1: a randomized placebo and active-controlled phase III study investigating oliceridine (TRV130), a G protein-biased ligand at the micro-opioid receptor, for management of moderate-to-severe acute pain following bunionectomy. J Pain Res. 2019 Mar 11;12:927-943. doi: 10.2147/JPR.S171013. eCollection 2019. PMID 30881102
- [Result] Bergese SD, Brzezinski M, Hammer GB, Beard TL, Pan PH, Mace SE, Berkowitz RD, Cochrane K, Wase L, Minkowitz HS, Habib AS. ATHENA: A Phase 3, Open-Label Study Of The Safety And Effectiveness Of Oliceridine (TRV130), A G-Protein Selective Agonist At The micro-Opioid Receptor, In Patients With Moderate To Severe Acute Pain Requiring Parenteral Opioid Therapy. J Pain Res. 2019 Nov 14;12:3113-3126. doi: 10.2147/JPR.S217563. eCollection 2019. PMID 31814753
- [Result] Chu F, Yao Y, Gao B, Huang M, Kong L. Incidence and risk factors for potential drug-drug interactions in outpatients receiving opioid analgesics. Expert Opin Drug Saf. 2025 Feb;24(2):167-175. doi: 10.1080/14740338.2024.2346101. Epub 2024 Apr 23. PMID 38641999
- [Result] Bjornnes AK, Lie I, Parry M, Falk R, Leegaard M, Rustoen T, Valeberg BT. Association between self-perceived pain sensitivity and pain intensity after cardiac surgery. J Pain Res. 2018 Aug 1;11:1425-1432. doi: 10.2147/JPR.S167524. eCollection 2018. PMID 30122973